CLINICAL TRIAL: NCT00766350
Title: A Randomized, Pilot Clinical Trial to Assess the Comparative Efficacy and Tolerability of Quetiapine XR Versus Amitriptyline for the Treatment of Patients With Fibromyalgia
Brief Title: Comparative Efficacy and Tolerability of Quetiapine XR and Amitriptyline in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: AstraZeneca (Industry); Hospital Clinico Universitario San Cecilio (Other)
Responsible Party: Principal Investigator, Elena Pita Calandre, Professor of Pharmacology, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443C00024
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; quetiapine; amitriptyline
MeSH Terms: conditions — Fibromyalgia | interventions — Amitriptyline; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- amitriptyline (Active Comparator)
  Interventions: Drug: amitriptyline
- quetiapine (Experimental)
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: amitriptyline — initial dose 10 mg/day, target dose: 25 mg/day, maximum dose: 75 mg/day, dosage form: tablets, duration: 16 weeks
  Other Names: Tryptizol
  Arms: amitriptyline
Drug: quetiapine — initial dose: 50 mg/day, target dose: 100 mg/day, maximum dose: 300 mg/day, dosage form:extended release tablets , duration: 16 weeks
  Other Names: Seroquel XR
  Arms: quetiapine

SUMMARY:
Quetiapine, a second generation antipsychotic, has shown beneficial activity on fibromyalgia symptomatology, administered as add-on treatment, in a sample of 35 patients. The purpose of the present study is to compare, in a controlled setting, the efficacy and the tolerability of quetiapine extended release with amitriptyline in the treatment of patients with fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 70 years.
2. Meeting American College of Rheumatology criteria for primary fibromyalgia: widespread aching pain in all four quadrants of the body and axial skeleton and greater than or equal to 11 of 18 tender points under digital palpation examination.
3. A FIQ total score (0 100) of 40 or greater
4. A score of 4 or greater on the average pain item of the BPI
5. Written informed consent
6. Female patients of childbearing potential must be using a reliable contraceptive method and have a negative urine human chorionic gonadotropin (HCG) test at enrolment.
7. Able to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Evidence of current traumatic injury, inflammatory rheumatic disease, or infectious or endocrine related joint disease.
2. A lifetime history of hypomania, mania, psychosis or dementia.
3. Current primary Axis I diagnosis other than major depressive disorder
4. Substance or alcohol dependence at enrolment and within the past 12 months (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM IV
5. Severe depression as evidenced by a Beck Depression Inventory score ≥ 30
6. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
7. History of seizures
8. Known lack of response to 2, or more than 2, different type of antidepressants in depression of fibromyalgia.
9. Pregnancy or breast feeding.
10. Patients with a history of urinary retention, angle closure glaucoma, or increased intraocular pressure.
11. Patients with known cardiovascular disease (history of myocardial infarction or ischemic heart disease, heart failure or conduction abnormalities), cerebrovascular disease or conditions which would predispose patients to severe hypotension (dehydration, hypovolemia and treatment with antihypertensive medications).
12. Patients who have received IMAOs, SSRIs or other antidepressants within two weeks of randomization.
13. Current or past history of kidney or liver insufficiency
14. Prior to randomization. Unwillingness to discontinue previously prescribed drugs for fibromyalgia other than those authorized in the protocol, as acetaminophen and bromazepam
15. Patients who have received quetiapine or amitriptyline within 1 year of randomization.
16. Patients with known intolerance or lack of response to quetiapine fumarate and/or amitriptyline, as judged by the investigator
17. Use of any of the following cytochrome P450 3A4 inhibitors within 14 days of enrolment, including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine, and saquinavir
18. Use of any of the following cytochrome P450 inducers within 14 days of enrolment, including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's wort, and glucocorticoids
19. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM IV criteria within 4 weeks of enrolment
20. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment, with clinical relevance.
21. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension), as judged by the investigator
22. Involvement in planning and conduct of the study
23. Previous enrolments or randomisation of treatment in the present study.
24. Participation in another trial with drugs within 4 weeks of enrolment into this study or a longer period in accordance with local requirements.
25. Patients with uncontrolled Diabetes Mellitus (DM)
26. An absolute neutrophil count (ANC) equal or lower than 1.5 x 109 per liter.
27. Patients who show at the randomization visit a reduction in the FIQ total score equal or greater than 20% from the screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to endpoint in the total score of Fibromyalgia Impact Questionnaire | baseline, 4, 8, 12 and 16 weeks

SECONDARY OUTCOMES:
Change from baseline to endpoint in the scores of the Brief Pain Inventory, the Pittsburgh Sleep Quality Inventory, the Beck Depression Inventory, and the State and Trait Anxiety Inventory | baseline, 4, 8, 12 and 16 weeks
Discontinuation rates due to treatment-related adverse events, proportion of patients experiencing adverse events, proportion of patients experiencing serious adverse events, adverse events description and classification. | baseline, 0, 4, 8, 12 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena P Calandre, MD, Principal Investigator — Clinical Pharmacology Department of the Hospital Clinico Universitario San Cecilio
Locations (1):
- Hospital Clinico Universitario San Cecilio, Granada, Granada, Spain

REFERENCES:
- [Background] Hidalgo J, Rico-Villademoros F, Calandre EP. An open-label study of quetiapine in the treatment of fibromyalgia. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jan 30;31(1):71-7. doi: 10.1016/j.pnpbp.2006.06.023. Epub 2006 Aug 4. PMID 16889882